CLINICAL TRIAL: NCT04753840
Title: Long-term of Remote Ischemic Preconditioning in Patients With Mild Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanICE202103
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Antihypertensive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental A: Drug group+lifestyle intervention (Experimental): Experimental group A used only one antihypertensive drug (ACEI / ARB, beta blocker, calcium channel blocker, diuretic, etc.) plus lifestyle intervention to control blood pressure.
  Interventions: Other: Antihypertensive drugs; Behavioral: lifestyle intervention
- Experimental B: RIPC group+lifestyle intervention (Experimental): The experimental group B received ripc treatment of upper limbs every day plus lifestyle intervention until the end of the follow-up. The treatment time was 40 minutes per day, 10 minutes as a cycle (cuff inflated to 200 mmHg and maintained for 5 minutes, then deflated for 5 minutes to start the next cycle), a total of 4 cycles.
  Interventions: Other: remote ischemic preconditioning（RIPC）; Behavioral: lifestyle intervention
- Experimental c: lifestyle intervention (Other): The control group take lifestyle intervention to control blood pressure, such as changing dietary habits, smoking cessation and alcohol restriction, exercise and so on.
  Interventions: Behavioral: lifestyle intervention

INTERVENTIONS:
Other: Antihypertensive drugs — One of ACEI / ARB, beta blocker, calcium channel blocker, diuretic
  Arms: Experimental A: Drug group+lifestyle intervention
Other: remote ischemic preconditioning（RIPC） — 40 minutes per day, 10 minutes as a cycle (cuff inflated to 200 mmHg and maintained for 5 minutes, then deflated for 5 minutes to start the next cycle)， a total of 4 cycles.
  Arms: Experimental B: RIPC group+lifestyle intervention
Behavioral: lifestyle intervention — Such as changing dietary habits, smoking cessation and alcohol restriction, exercise and so on.

SUMMARY:
According to the latest survey data of China hypertension annual meeting, there are about 300 million patients with hypertension in China, with 10 million new cases of hypertension each year, and there is an obvious trend of younger people. In particular, young and middle-aged people are in a state of mild hypertension for a long time, which causes great pressure on health and medical treatment. At present, the main clinical measures for mild hypertension are to change their eating habits, quit smoking and alcohol, exercise and other lifestyle changes, as well as drug control. For most patients with mild hypertension, drug control is not the best choice. It has been reported that remote ischemic preconditioning (RIPC) may play an effective role in reducing blood pressure .The purpose of this study was to investigate the extent of long-term application of RIPC to reduce blood pressure in patients with mild hypertension.

DETAILED DESCRIPTION:
A total of 200 patients with mild hypertension were enrolled in this study, using the method of open label and parallel grouping; 100 cases in the experimental group and 100 cases in the control group, The experimental group was divided into life intervention + drug group and life intervention + ripc group, with 50 patients in each group. The results of 24-hour ambulatory blood pressure monitoring (ABPM) of the three groups were observed before and 3 months after use, including HR, pulse pressure, 24-hour systolic blood pressure, 24-hour diastolic blood pressure, daytime systolic blood pressure, daytime diastolic blood pressure, nighttime systolic blood pressure and nighttime diastolic blood pressure. The changes of renalase, catecholamine, renin, angiotensin - Ⅱ, aldosterone, RhoA kinase, no, adenosine and bradykinin were observed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed patients with mild hypertension (SBP: 140~159mmHg; DBP: 90~99mmHg)

Exclusion Criteria:

* Cannot tolerate RIPC
* Non-essential hypertension
* patients who have uncontrolled severe arrhythmia, diabetes, electrolyte disturbance
* patients who have severe organic diseases such acute myocardial infarction, cardiac insufficiency, abnormal renal function, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-07-03 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean systolic blood pressure | 3 months
  24-hour Mean systolic blood pressure measured by Ambulatory blood pressure monitoring
Mean diastolic blood pressure | 3 months
  24-hour Mean diastolic blood pressure measured by Ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Concentration of Renalase | 3 months
  blood renalase concentration
Concentration of catecholamine | 3 months
  Blood catecholamine concentration
Concentration of adenosine | 3 months
  blood adenosine concentration
Concentration of bradykinin | 3 months
  blood bradykinin concentration
Concentration of renin | 3 months
  blood renin concentration

CONTACTS AND LOCATIONS:
Overall Officials: Muwei Li, MD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai central China Cardiovascular hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
IPD can be obtained from the researcher upon reasonable request

REFERENCES:
- [Background] Jones H, Hopkins N, Bailey TG, Green DJ, Cable NT, Thijssen DH. Seven-day remote ischemic preconditioning improves local and systemic endothelial function and microcirculation in healthy humans. Am J Hypertens. 2014 Jul;27(7):918-25. doi: 10.1093/ajh/hpu004. Epub 2014 Mar 13. PMID 24627443
- [Background] Moro L, Pedone C, Mondi A, Nunziata E, Antonelli Incalzi R. Effect of local and remote ischemic preconditioning on endothelial function in young people and healthy or hypertensive elderly people. Atherosclerosis. 2011 Dec;219(2):750-2. doi: 10.1016/j.atherosclerosis.2011.08.046. Epub 2011 Sep 7. PMID 21945497